CLINICAL TRIAL: NCT01404455
Title: Effect of Wide Pulse Pressure on the Predictability of Stroke Volume Variation for Fluid Responsiveness in Patients Undergoing Off-pump Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, MD, PhD, Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB 1-2010-0039
Record Dates: First submitted 2011-04-01; First posted 2011-07-28 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Stroke Volume Variation
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Normal pulse pressure (Other): pulse pressure <60mmHg
  Interventions: Other: HES 130/0.4 (VoluvenⓇ, Fresenius Kabi, Graz, Austria) 500mL loading
- Wide pulse pressure (Other): pulse pressure ≥60mmHg
  Interventions: Other: HES 130/0.4 (VoluvenⓇ, Fresenius Kabi, Graz, Austria) 500mL loading

INTERVENTIONS:
Other: HES 130/0.4 (VoluvenⓇ, Fresenius Kabi, Graz, Austria) 500mL loading — HES 130/0.4 (VoluvenⓇ, Fresenius Kabi, Graz, Austria) 500mL loading during 15 minutes after induction of anesthesia

SUMMARY:
The investigators examined the predictability of stroke volume variation for fluid responsiveness in patients with wide pulse pressure undergoing off-pump coronary artery bypass graft

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 20
* 2. elective off-pump coronary artery bypass graft

Exclusion Criteria:

* 1. arrhythmia
* 2.EF <40%
* 3.valvular heart dz
* 4.pul HTN
* 5.PAOD
* 6.lung dz
* 7.NYHA IV
* 8.ESRD

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The predictability of stroke volume variation for fluid responsiveness in patients with wide pulse pressure | 30 min

SECONDARY OUTCOMES:
Cut off value of stroke volume variation for predicting fluid responsiveness in patients with wide pulse pressure | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea